CLINICAL TRIAL: NCT07074470
Title: A Prospective Study of Combination Regimen of Teniposide, PD-1 Monoclonal Antibody and Selinixor for Patients With Relapsed and Refractory Primary Central Nervous System Lymphoma.
Brief Title: Combination Regimen of Teniposide, PD-1 Monoclonal Antibody and Selinixor for Patients With Relapsed or Refractory PCNSL
Acronym: VPX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024474
Record Dates: First submitted 2025-07-09; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Primary Central Nervous System Lymphoma (PCNSL)
Keywords: VPX; PCNSL; teniposide; PD-1; selinexor
MeSH Terms: interventions — Teniposide; Thiotepa; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (ASCT-eligible) (Experimental): Patients achieving response after 2 cycles of VPX regimen will proceed to ASCT as consolidation therapy followed by PD-1 monoclonal antibody therapy maintenance for up to 2 years, or until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: Induction therapy-2 cycles of VPX (Teniposide, PD-1 monoclonal antibody plus Selinixor); Procedure: Consolidation therapy with ASCT after TB (Thiotepa plus Busulfan) preconditioning; Drug: Maintenance treatment-PD-1 monoclonal antibody
- Cohort 2 (ASCT-ineligible) (Experimental): Patients achieving response after 2 cycles of VPX regimen will receive four additional cycles of VPX regimen, followed by whole-brain radiotherapy (WBRT) consolidation. After consolidation therapy, patients will receive PD-1 monoclonal antibody maintenance therapy for up to 2 years, or until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: Induction therapy-2 cycles of VPX (Teniposide, PD-1 monoclonal antibody plus Selinixor); Drug: Consolidation therapy-4 cycles of VPX (Teniposide, PD-1 monoclonal antibody plus Selinixor); Radiation: Consolidation therapy-whole brain radiation therapy; Drug: Maintenance treatment-PD-1 monoclonal antibody

INTERVENTIONS:
Drug: Induction therapy-2 cycles of VPX (Teniposide, PD-1 monoclonal antibody plus Selinixor) — 2 cycles of VPX regimen (21days per cycle) Teniposide: intravenous drip, 50mg d1-3; PD-1 monoclonal antibody: intravenous drip, 200mg d1; Selinixor: take 40mg orally, W1，60mg，W2，40mg biw，W3，cycle 1； 40mg， biw，cycle 2
Procedure: Consolidation therapy with ASCT after TB (Thiotepa plus Busulfan) preconditioning — TB preconditioning:
  Thiotepa intravenous drip 300mg/m2 d-6-d-5; Busulfan: intravenous drip, 0.8mg/kg q6h d-4--d2; followed by autologous peripheral stem cells infusion at day 0
  Arms: Cohort 1 (ASCT-eligible)
Drug: Consolidation therapy-4 cycles of VPX (Teniposide, PD-1 monoclonal antibody plus Selinixor) — 4 cycles of VPX regimen (21days per cycle) Teniposide: intravenous drip, 50mg d1-3; PD-1 monoclonal antibody: intravenous drip, 200mg d1; Selinixor: take 40mg orally biw, cycle 3-6；
  Arms: Cohort 2 (ASCT-ineligible)
Radiation: Consolidation therapy-whole brain radiation therapy — whole brain radiotherapy: CTV1: 20-30Gy/10fractions GTVp: 25-40Gy/10fractions
  Arms: Cohort 2 (ASCT-ineligible)
Drug: Maintenance treatment-PD-1 monoclonal antibody — PD-1 monoclonal antibody for up to 2 years intravenous infusion, 200mg d1 (21days per cycle)

SUMMARY:
This study aims to evaluate the efficacy and safety of the VPX regimen, a novel combination of teniposide, PD-1 monoclonal antibody and selinexor, in patients with relapsed/refractory (R/R) primary central nervous system lymphoma (PCNSL) who have progressed after high-dose methotrexate (HD-MTX)-based systemic therapy. By investigating this therapeutic approach, we seek to establish a new treatment paradigm that may improve clinical outcomes of this high-risk population.

DETAILED DESCRIPTION:
This study will enroll patients aged 18-75 years with R/R PCNSL who have progressed after HD-MTX-based systemic therapy. Eligible participants will receive induction therapy with 2 cycles of VPX regimen followed by evaluation of contrast-enhanced magnetic resonance imaging (MRI) of the brain. Patients who got disease progression of stable disease will be withdrawn from this study. Patients who achieved partial remission(PR) or complete remission（CR）will receive consolidation treatment stratification as followings:

Group A (ASCT-eligible): Patients will proceed to autologous stem cell transplantation (ASCT) as consolidation therapy.

Group B (ASCT-ineligible): Patients will receive four additional cycles of VPX regimen, followed by whole-brain radiotherapy (WBRT) consolidation.

After consolidation therapy, all responders will receive PD-1 monoclonal antibody therapy maintenance for up to 2 years, or until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old (inclusive).
2. Participants must be able to understand and willing to sign a written informed consent form.
3. The Eastern Cooperative Oncology Group is in a state of 0 to 3.
4. The expected lifespan is ≥ 3 months (according to researchers).
5. Primary central nervous system lymphoma of B-cell origin confirmed by pathology (histology or cytology).
6. Measurable diseases are defined as having a short diameter of at least 1.0cm through enhanced MRI.
7. Recurrent/refractory PCNSL: Must have received at least one systemic treatment based on high-dose methotrexate.
8. Any non hematological toxicity related to previous treatment should be restored to grade 1 or normal (excluding hair loss according to NCI CTCAE 5.0).
9. Bone marrow and organ function meet the following criteria (no blood transfusion, no G-CSF, no medication correction within 14 days prior to screening):

   Bone marrow function: absolute value of neutrophils ≥ 1.5 × 10 ^ 9/L, platelets ≥ 80 × 10 ^ 9/L, hemoglobin ≥ 80 g/L; Liver function: serum total bilirubin ≤ 1.5 × ULN (≤ 3.0 × ULN, if there is liver metastasis); Glutamate oxalate transaminase (AST) and glutamate pyruvate transaminase (ALT) ≤ 2.5 × ULN (≤ 5.0 × ULN, if there is liver metastasis); Coagulation function: International normalized ratio (INR) and activated partial thromboplastin time ≤ 1.5 × ULN; Renal function: serum creatinine ≤ 1.5 × ULN or estimated creatinine clearance rate ≥ 60 mL/min (male: Cr (ml/min)=(140 years old) × body weight (kg)/72 × serum creatinine concentration (mg/dl); Female: Cr (ml/min)=(140 years old) x body weight (kg)/85 x serum creatinine concentration (mg/dl)
10. Women with reproductive potential must agree to use efficient contraceptive methods during treatment and within 6 months after the last study drug administration. Sexually active males must agree to use highly effective contraceptive measures during treatment and within 6 months after the last dose of medication.
11. Can accept multiple MRI/CT and lumbar puncture examinations.
12. Swallowing oral tablets/capsules is not difficult.
13. Good compliance, willing to follow inspection procedures such as visit schedule, medication schedule, laboratory tests, etc.

Exclusion Criteria:

1. Chemotherapy, radiotherapy, immunotherapy, or antibody therapy for anti-tumor treatment, or herbal medicine with anti-tumor indications, small molecule targeted therapy within 2 weeks, monoclonal antibody conjugate drug or cytotoxic therapy within 10 weeks.
2. Participate in another clinical study using the research product within 4 weeks prior to the first day of treatment.
3. Patients who have used systemic corticosteroids for more than 5 days within 14 days prior to medication or require daily administration of>10mg dexamethasone or equivalent medication to control central nervous system disorders.
4. Active concurrent malignant tumors that require active treatment.
5. Patients who have received previous treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, selenidazole, and tiniposide drugs within 6 months prior to initial administration.
6. Suffering from uncontrolled or severe cardiovascular disease, including (but not limited to): any of the following: congestive heart failure (NYHA class III or IV); miocardial infarction; Unstable angina pectoris; Or there may be arrhythmia requiring treatment during screening, and the left ventricular ejection fraction (LVEF) within 6 months prior to initial administration is less than 50%; Primary cardiomyopathy (e.g. dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, undefined cardiomyopathy); A clinically significant medical history of QTc prolongation, grade II type II atrioventricular block or grade III atrioventricular block, or QTc interval (Method F)>470 milliseconds (females) or>480 milliseconds (males); Atrial fibrillation (EHRA ≥ 2b); Uncontrollable hypertensive patients are considered unsuitable to participate in this study.
7. Uncontrolled infections or infections requiring intravenous antibiotic treatment.
8. Chronic hepatitis B carriers with active hepatitis B or C infection (hepatitis B: acute hepatitis B, untreated chronic hepatitis B virus infection, HBV-DNA ≥ detection limit of each center; hepatitis C: HCV RNA positive) or syphilis. Attention: Non active carriers of HBV surface antigen (HBsAg), active HBV infection and persistent anti HBV suppression (HBV DNA<detection limit per center) subjects, as well as HCV cured subjects, can be recruited.

   Human immunodeficiency virus (HIV) infection
9. Clinically significant gastrointestinal abnormalities that may affect drug intake, transportation, or absorption (such as active gastrointestinal inflammation, chronic diarrhea, intestinal obstruction, etc.), or total gastrectomy or gastric banding surgery.
10. Previous allogeneic stem cell transplantation. Or those who have the intention of allogeneic hematopoietic stem cell transplantation;
11. For female participants, they are currently pregnant or breastfeeding.
12. Allergic to research drugs or excipients.
13. The patient has active mental illness, alcohol, drug or substance abuse.
14. There are any life-threatening diseases, medical conditions, or organ system dysfunction that researchers believe may affect patient safety or compliance with research procedures.
15. There are other researchers who believe that it is not suitable to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2030-01-02 (Estimated); Study Completion 2032-01-02 (Estimated)

PRIMARY OUTCOMES:
Overall response rate(ORR) | At the end of 2 cycles of VPX regimen (each cycle is 21 days)
  The rate of patients who achieved CR or PR after induction therapy with 2 cycles of VPX regimen

SECONDARY OUTCOMES:
2-year progression-free survival(PFS) | From enrollment to 2-year after the end of last patient's treatment
  PFS will be assessed from the first day of treatment to date of progression, relapse, death or end of follow-up.
Major adverse events | From enrollment to 1 month after induction therapy
  The safety and tolerability of the VPX regimen measured by the major adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kasamon YL, Price LSL, Okusanya OO, Richardson NC, Li RJ, Ma L, Wu YT, Theoret M, Pazdur R, Gormley NJ. FDA Approval Summary: Selinexor for Relapsed or Refractory Diffuse Large B-Cell Lymphoma. Oncologist. 2021 Oct;26(10):879-886. doi: 10.1002/onco.13859. Epub 2021 Jul 1. PMID 34132444
- [Background] Houillier C, Dureau S, Taillandier L, Houot R, Chinot O, Molucon-Chabrot C, Schmitt A, Gressin R, Choquet S, Damaj G, Peyrade F, Abraham J, Delwail V, Gyan E, Sanhes L, Cornillon J, Garidi R, Delmer A, Al Jijakli A, Morel P, Waultier A, Paillassa J, Chauchet A, Gastinne T, Laadhari M, Plissonnier AS, Feuvret L, Cassoux N, Touitou V, Ricard D, Hoang-Xuan K, Soussain C; LOC Network for CNS Lymphoma. Radiotherapy or Autologous Stem-Cell Transplantation for Primary CNS Lymphoma in Patients Age 60 Years and Younger: Long-Term Results of the Randomized Phase II PRECIS Study. J Clin Oncol. 2022 Nov 10;40(32):3692-3698. doi: 10.1200/JCO.22.00491. Epub 2022 Jul 14. PMID 35834762